CLINICAL TRIAL: NCT02098746
Title: Sonias Combination Tablets LD Special Drug Use Surveillance Survey in Patients With Type 2 Diabetes Mellitus Who Respond Poorly to Pioglitazone
Brief Title: Pioglitazone/Glimepiride (Sonias) Combination Tablets Special Drug Use Surveillance Survey in Patients With Type 2 Diabetes Mellitus Who Respond Poorly to Pioglitazone
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 097-012; JapicCTI-142445 (Registry Identifier: JapicCTI); JapicCTI-R150762 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes
Keywords: Pharmacological therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; glimepiride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pioglitazone/glimepiride: Pioglitazone/glimepiride 15 mg/1 mg, orally once daily before or after breakfast.
  Interventions: Drug: Pioglitazone/glimepiride

INTERVENTIONS:
Drug: Pioglitazone/glimepiride — Pioglitazone/glimepiride combination tablets
  Other Names: Sonias combination tablets LD

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of long-term use of pioglitazone/glimepiride combination tablets (Sonias Combination Tablets LD) in patients with type 2 diabetes mellitus who respond poorly to pioglitazone hydrochloride monotherapy (pioglitazone at 15 mg/day) in the routine clinical setting.

DETAILED DESCRIPTION:
This is a special drug use surveillance on long-term use of pioglitazone/glimepiride combination tablets (Sonias Combination Tablets LD) designed to investigate the frequency of adverse drug reactions in patients with type 2 diabetes mellitus who respond poorly to pioglitazone hydrochloride monotherapy (pioglitazone at 15 mg/day).

The usual adult dosage is one tablet (15 mg/1 mg of pioglitazone/glimepiride) administered orally once daily before or after breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus for whom treatment with pioglitazone hydrochloride monotherapy (pioglitazone at 15 mg/day) is considered inefficacious as per physician's assessment and for whom long-term treatment with pioglitazone/glimepiride combination tablets is considered necessary

Exclusion Criteria:

* (1) Patients with cardiac failure or a history of cardiac failure (2) Patients with serious hepatic or renal impairment (3) Patients with severe ketosis, diabetic coma or precoma, or type 1 diabetes mellitus (4) Patients with severe infection, severe trauma, or pre- and post-operative patients (5) Patients with gastrointestinal disorders such as diarrhea and vomiting (6) Pregnant or potentially pregnant women (7) Patients with a history of hypersensitivity to the ingredients in Sonias Combination Tablets or sulfonamides

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2011-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This observational study took part at 64 investigative sites in Japan from 15 June 2011 to 31 July 2014.
Pre-assignment Details: Participants with a diagnosis of type 2 diabetes mellitus receiving treatment with pioglitazone/glimepiride 15 mg/1 mg once daily in routine clinical practice, because pioglitazone alone was not considered effective, were enrolled in the study.
Period: Overall Study
Arm/Group | Pioglitazone/Glimepiride
Started | 294
Completed | 289
Not Completed | 5
Not completed — Changes of Investigator | 2
Not completed — Other Miscellaneous Reasons | 1
Not completed — Enrolled 15 Days After the First Dose | 1
Not completed — Data Not Available After Treatment | 1

BASELINE CHARACTERISTICS:
Population: Baseline measures are based on the Safety Analysis Set (safety assessment population) that included all patients who received at least one dose of pioglitazone/glimepiride.
Arm/Group | Pioglitazone/Glimepiride
Number analyzed (Participants) | 289
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (12.56)
Age, Customized [Number; unit: participants]
  <65 years | 112
  ≥65 years | 177
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117
  Male | 172
Pregnancy Status (Females Only) [Number; unit: participants] — Data based on female participants only (N=117).
  participants
    Not pregnant | 117
    Pregnant | 0
Duration of Type 2 Diabetes [Mean (Standard Deviation); unit: years] — Duration of type 2 diabetes data was available for 207 participants.
  years | 6.19 (5.444)
Duration of Type 2 Diabetes, Categorical [Number; unit: participants]
  <2 years | 56
  ≥2 to <5 years | 44
  ≥5 to <10 years | 58
  ≥10 years | 49
  Unknown | 82
Categories of Health Care [Number; unit: participants]
  Outpatient | 287
  Inpatient | 2
History of Allergy [Number; unit: participants]
  No | 239
  Yes | 29
  Unknown | 21
Complications of Type 2 Diabetes [Number; unit: participants]
  No | 25
  Yes | 264
Breakdown of Complications (Tabulated in Duplicate) [Number; unit: participants] — Tabulated in duplicate = participants may be accounted for in more than one category.
  participants
    Microangiopathy | 31
    Diabetic nephropathy | 17
    Diabetic retinopathy | 9
    Diabetic neuropathy | 12
    Hypertension | 175
    Dyslipidaemia | 175
    Hyperuricaemia | 29
    Liver disease | 25
    Renal disease | 18
    Heart disease | 17
    Cerebrovascular disease | 15
    Malignant tumor | 1
    Other | 12
Presence of Medical History [Number; unit: participants]
  No | 228
  Yes | 39
  Unknown | 22
Weight [Mean (Standard Deviation); unit: kg] — Weight data was available for 250 participants.
  kg | 65.64 (13.662)
Weight, Categorical [Number; unit: participants]
  <40 kg | 1
  ≥40 to <50 kg | 24
  ≥50 to <60 kg | 57
  ≥60 to <70 kg | 81
  ≥70 kg | 87
  Unmeasured | 39
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI data was available for 242 participants.
  kg/m^2 | 25.45 (4.230)
BMI, Categorical [Number; unit: participants]
  <18.5 kg/m^2 | 8
  ≥18.5 to <25 kg/m^2 | 107
  ≥25 to <30 kg/m^2 | 97
  ≥30 kg/m^2 | 30
  Unknown | 47
History of Alcohol (Drinking Alcohol-Containing Beverages Nearly Every Day) [Number; unit: participants]
  Yes | 167
  No | 81
  Unknown | 41
Smoking Classification [Number; unit: participants]
  Never Smoked | 134
  Current Smoker | 54
  Ex-smoker | 55
  Unknown | 46
Compliance Rate with the Diet Regimen (at the Start of Treatment with Sonias Combination Tablets LD) [Number; unit: participants]
  ≥ 90% | 73
  ≥ 70% | 118
  ≥ 50% | 53
  < 50% | 18
  Not performed or compliance status is unknown | 27
Compliance Rate with the Exercise Regimen (at Start of Treatment with Sonias Combination Tablets LD) [Number; unit: participants]
  ≥ 90% | 49
  ≥ 70% | 97
  ≥ 50% | 76
  < 50% | 36
  Not performed or compliance status is unknown | 31
Glycosylated hemoglobin A1c (HbA1c) (at Start of Treatment with Sonias Combination Tablets LD) [Mean (Standard Deviation); unit: %] — HbA1c data was available for 264 participants.
  % | 7.75 (1.493)
HbA1c, Categorical [Number; unit: participants]
  < 6.0% | 8
  ≥ 6.0% to < 7.0% | 66
  ≥ 7.0% to < 8.0% | 110
  ≥ 8.0% | 80
  Unknown | 25

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Drug Reactions
Description: Frequency of adverse drug reactions is defined as the number of participants with adverse drug reactions. Frequency, seriousness, and time to onset of adverse drug reactions were tabulated by each symptom. Adverse events are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug. Among these, events which are considered possibly associated with a medicinal product are defined as adverse drug reactions.
Time Frame: 12 months
Population: The Safety Analysis Set (safety assessment population) included all patients who received at least one dose of pioglitazone/glimepiride (N=289).
Measure: Number; unit: participants
Arm/Group | Pioglitazone/Glimepiride
Number analyzed (Participants) | 289
participants
  Anaemia | 1
  Hypoglycaemia | 7
  Generalised oedema | 1
  Oedema | 1
  Weight increased | 6

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: Tabulation of HbA1c values and the changes from Baseline at each test time point (test value at each test time point after Baseline - test value at Baseline). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Months 3, 6, 9, 12 and at Final assessment
Population: The analysis was performed on the efficacy assessment population (N=250) with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Pioglitazone/Glimepiride
Number analyzed (Participants) | 250
percent
  Month 3 (n=234) | -0.83 (1.030)
  Month 6 (n=190) | -0.84 (1.094)
  Month 9 (n=177) | -0.83 (1.088)
  Month 12 (n=84) | -0.62 (1.139)
  Final Assessment (n=247) | -0.92 (1.285)

3. Secondary Outcome: Change From Baseline in Fasting Blood Glucose Level
Description: Tabulation of fasting blood glucose level and the changes from Baseline at each test time point (test value at each test time point after Baseline - test value at Baseline). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Months 3, 6, 9, 12 and at Final assessment
Population: The analysis was performed on the efficacy assessment population (N=250) with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pioglitazone/Glimepiride
Number analyzed (Participants) | 250
mg/dL
  Month 3 (n=76) | -15.9 (35.99)
  Month 6 (n=59) | -23.2 (40.11)
  Month 9 (n=53) | -12.7 (37.60)
  Month 12 (n=28) | -17.0 (20.42)
  Final Assessment (n=83) | -17.7 (42.23)

4. Secondary Outcome: Change From Baseline in Fasting Insulin Level
Description: Tabulation of fasting insulin level and the changes from Baseline at each test time point (test value at each test time point after Baseline - test value at Baseline). A negative change from Baseline indicates improvement. A positive change from Baseline indicates a worsening.
Time Frame: Baseline, Months 3, 6, 9, 12 and at Final assessment
Population: The analysis was performed on the efficacy assessment population (N=250) with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: μU/dL
Arm/Group | Pioglitazone/Glimepiride
Number analyzed (Participants) | 250
μU/dL
  Month 3 (n=33) | 1.66 (9.419)
  Month 6 (n=25) | -0.25 (3.976)
  Month 9 (n=17) | 1.32 (3.949)
  Month 12 (n=15) | -0.29 (3.489)
  Final Assessment (n=39) | 0.98 (7.310)

5. Primary Outcome: Frequency of Serious Adverse Drug Reactions
Description: Frequency of serious adverse drug reactions is defined at the number of participants with serious adverse drug reactions. Frequency of serious adverse drug reactions were tabulated by each symptom. Adverse events are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug. A serious adverse event is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant. Among these, events which are considered possibly associated with a medicinal product are defined as adverse drug reactions.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pioglitazone/Glimepiride
Number analyzed (Participants) | 289
participants | 0

ADVERSE EVENTS:
Time Frame: 12 Months
Description: Safety Analysis Set included all patients who received at least one dose of pioglitazone/glimepiride. At each visit the investigator documented any occurrence of adverse events. Any event that occurred during the observation period was recorded, irrespective of the relation to study treatment.
Arm/Group | Pioglitazone/Glimepiride
Serious Adverse Events (participants affected / at risk) | 2/289
Other Adverse Events (participants affected / at risk) | 0/289
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone/Glimepiride (N=289)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Atrioventricular block complete (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.